CLINICAL TRIAL: NCT03262350
Title: Can Yoga Reduce Body Image Concerns in Females, Thereby Reducing Risk of Obesity and Eating Disorders?
Brief Title: The Effects of Yoga on Body Image in College Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: University of Minnesota (Other); The Emily Program (Unknown); Neuropsychiatric Research Institute (Unknown)
Responsible Party: Principal Investigator, Carly R Pacanowski, Assistant Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REF AWARD# 0001271422
Record Dates: First submitted 2017-05-01; First posted 2017-08-25 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Body Image; Eating Disorder; Obesity; Yoga
MeSH Terms: conditions — Feeding and Eating Disorders; Obesity | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): Participants are required to attend three assessment visits. During these assessments, participants will complete a questionnaire that will ask about their eating patterns, body image, sleep habits, and loneliness and have their height and weight measured. Participants are also required to attend 50-minute yoga classes on Mondays, Wednesdays, and Fridays from 1:25-2:15pm for 10 weeks. The overall time commitment for Yoga Group participants is 3 hours of assessments and 50-minute yoga classes 3X week for 10 weeks.
  Interventions: Behavioral: Yoga
- Control Group (No Intervention): Participants will be required to attend three assessment visits. During these assessments, participants will complete a questionnaire that will ask about their eating patterns, health habits, body image, sleep habits and loneliness and have their height and weight measured. The overall time commitment for Control Group participants is 3 hours of assessments total.

INTERVENTIONS:
Behavioral: Yoga — The yoga classes will be adapted to all levels of experience, mobility, and body size. Specific breathing techniques and body positive language will be incorporated into a body-positive yoga training done by Ms. Lisa Diers, RDN, E-RYT, YACEP. Less focus will be placed on precision of the poses, instead focus will be on body feelings, except where physically dangerous. Thus, the overall focus will be on listening to one's own body. List of messages will be carefully designed to be related to eating and weight, but to not be directly discussed. Ms. Diers will travel to Delaware to lead the intervention training for yoga instructors prior to the study taking place.
  Arms: Yoga Group

SUMMARY:
The purpose of this study is to assess the effects of a regular yoga practice on body image in college women.

DETAILED DESCRIPTION:
A randomized controlled design will be used to study the effects of a regular yoga practice on body image in young adult women. Fifty female freshman, sophomores, and juniors between the ages of 18 and 26 years will be recruited from the University of Delaware student population, specifically targeting those new to yoga. Age, academic standing, availability and prior yoga experience will be evaluated.

Consented individuals will be randomized to one of two conditions: (1) yoga (offered 3 times per week) for 10 weeks; or (2) a control group. Baseline assessments, midpoint assessments, and end-of-study assessments will be conducted on all participants. Participants will be compensated for their attendance at assessment visits.

ELIGIBILITY:
Inclusion Criteria:

* Freshman, sophomore, or junior at the University of Delaware
* Available Spring 2017 on Mondays, Wednesdays, and Fridays from 1:25-2:15pm
* Physically able to participate in yoga

Exclusion Criteria:

* Females who are seniors at the University of Delaware (This is because participants in the control condition will be given a pass to participate in group fitness at the end of the study, and would not be able to use this incentive if they are seniors)

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Body Image | 10 weeks
  assessed using Body Image Quality of Life Inventory
body image | 10 weeks
  assessed using Mind Body Self Relations Questionnaire

SECONDARY OUTCOMES:
change in Body Mass Index | 10 weeks
  weight and height will be combined to report BMI in kg/m^2
disordered eating attitudes/behaviors | 10 weeks
  assessed using the Eating Attitudes Test-26
disordered eating attitudes/behaviors | 10 weeks
  assessed using the Binge Eating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No